CLINICAL TRIAL: NCT05312073
Title: Study of In Vivo and in Vitro Transcriptomic and Proteomic Signatures in Unhereditary Ichtyosis
Acronym: OMICHTYOSE
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: APHP210692
Record Dates: First submitted 2021-12-10; First posted 2022-04-05 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Autosomal Recessive Congenital Ichthyosis; Epidermolytic Ichthyosis
MeSH Terms: conditions — Hyperkeratosis, Epidermolytic

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Patients with ichtyosis (Other)
  Interventions: Other: Biological samples
- Patients without ichtyosis (Other)
  Interventions: Other: Skin biopsy

INTERVENTIONS:
Other: Biological samples — Blood samples Superficial skin Biopsy Collection of fallen squames Tapes - stripping
  Arms: Patients with ichtyosis
Other: Skin biopsy — healthy skin from surgery interventions
  Arms: Patients without ichtyosis

SUMMARY:
The goal of this study is to identify important biological pathways involved in a variety of ichtyosis, using transcriptomic and proteomic techniques, with the aim of guiding the development of new therapeutis.

ELIGIBILITY:
Inclusion Criteria:

* Aged 15-80 years old
* Having an ARCI or EI, confirmed by a molecular diagnosis of a mutation in at least one of the following genes: TGM1, ALOX12B, NIPAL4, ABCA12, keratin 1 and keratin 10)
* Having stopped all topical treatments in at least 1% of the total body surface (equivalent to one palm of the hand of the patient), at least 8 days before the skin biopsy (which will be performed on this untreated area).
* Patients having a molecular diagnostic of genetic ichtyosis
* No contraindication to skin biopsy
* Health insurance coverage
* Signature of written consent

Exclusion Criteria:

* Aged less than 15 of over 80 years old
* Ichtyosis without a molecular confirmed diagnosis or with a different diagnosis
* History, in the 8 previous days, of any topical treatment on the area intended for the skin biopsy.
* No health insurance coverage
* Pregnant or breastfeeding woman
* Patient under guardianship or curatorship
* Patient under State Medical Assistance (AME)

Ages: 15 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-12-07 (Actual); Primary Completion 2024-04-06 (Actual); Study Completion 2024-04-06 (Actual)

PRIMARY OUTCOMES:
Transcript and protein levels of all genes measured by NGS mRNA sequencing and by mass spectrometry in lesioned skin biopsies | Up to 6 months post inclusion
  A two-fold increase or decrease in the transcript or protein levels between patients with different ARCI, EI, and between ARCI and EI patients and healthy controls (patients without ichtyosis) will allow to identify "upregulated" and "downregulated" genes.

SECONDARY OUTCOMES:
Transcript and protein levels of all genes assessed by NGS mRNA sequencing and by mass spectrometry (keratinocytes) | Up to 6 months post inclusion
  To determine, in vitro, the contribution from ARCI and EI keratinocytes in the overall transcriptomic and proteomic signature observed in vivo. A two-fold increase or decrease in the transcript or protein levels between patients and controls (th different ARCI, EI, and between ARCI and EI patients and healthy controls (patients without ichtyosis) will allow to identify "upregulated" and "downregulated" genes.
Phenotype of circulating PBMCS assessed by flow cytometry analysis using monoclonal Antibodies (mAbs) | Up to 6 months post inclusion

CONTACTS AND LOCATIONS:
Locations (1):
- Saint Louis Hospital, Paris, France

IPD SHARING:
Plan to Share IPD: Undecided